CLINICAL TRIAL: NCT01013753
Title: A Randomised, Double-Blind, Placebo- and Active-Controlled, Incomplete Crossover Efficacy and Safety Comparison of 4-week Treatment Periods of Once Daily Treatment of 4 Doses of BI 1744 CL Inhalation Solution Delivered by the Respimat® in Patients With Asthma
Brief Title: A Study of the Safety and Efficacy of 4 Doses of BI 1744 CL Delivered Via the Respimat in Patients With Asthma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1222.27; 2009-013395-48 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — olodaterol; Culture Media; Formoterol Fumarate

ARMS (6):
- Olodaterol (BI 1744) low (Experimental): Low dose inhaled orally once daily from the Respimat inhaler
  Interventions: Drug: Olodaterol (BI 1744) low
- Olodaterol (BI 1744) very low (Experimental): Very low dose inhaled orally once daily from the Respimat inhaler
  Interventions: Drug: Olodaterol (BI 1744) very low
- Olodaterol (BI 1744) medium (Experimental): Medium dose inhaled orally once daily from the Respimat inhaler
  Interventions: Drug: Olodaterol (BI 1744) medium
- Olodaterol (BI 1744) high (Experimental): High dose inhaled orally once daily from the Respimat inhaler
  Interventions: Drug: Olodaterol (BI 1744) high
- Formoterol 12 mcg (Active Comparator): 12mcg inhaled twice daily from the Aerolizer inhaler
  Interventions: Drug: Formoterol 12 mcg
- Placebo (Placebo Comparator): Olodaterol (BI 1744) placebo inhaled once daily from the Respimat inhaler and/or Formoterol placebo inhaled twice daily from the Aerolizer inhaler
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Determine efficacy and safety of Placebo inhaled once daily from the Respimat inhaler and/or twice daily from the Aerolizer inhaler
  Arms: Placebo
Drug: Olodaterol (BI 1744) high — Determine efficacy and safety in 4 different doses of Olodaterol (BI 1744) inhaled once daily via the Respimat
  Arms: Olodaterol (BI 1744) high
Drug: Olodaterol (BI 1744) medium — Determination of efficacy in 4 different doses of Olodaterol (BI 1744) inhaled once daily via the Respimat
  Arms: Olodaterol (BI 1744) medium
Drug: Olodaterol (BI 1744) very low — Determination of efficacy in 4 different doses of Olodaterol (BI 1744) inhaled once daily via the Respimat
  Arms: Olodaterol (BI 1744) very low
Drug: Formoterol 12 mcg — Determine efficacy and safety of 12 mcg Formoterol dose inhaled orally twice daily from the Aerolizer in comparison to other treatment groups
  Arms: Formoterol 12 mcg
Drug: Olodaterol (BI 1744) low — Determine efficacy and safety of 4 different doses of Olodaterol (BI 1744) inhaled once daily via the Respimat
  Arms: Olodaterol (BI 1744) low

SUMMARY:
The primary objective of this study is to determine the efficacy and safety of 4 doses of BI 1744 CL inhalation solution delivered by the Respimat® inhaler once daily for four weeks in patients with asthma in comparison to placebo.

ELIGIBILITY:
Inclusion criteria:

1. All patients must sign an informed consent consistent with International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) guidelines prior to participation in the trial, i.e. prior to any study procedures which includes medication washout and restrictions. A separate informed consent is required for pharmacogenomic sampling.
2. Male or female patients, aged between 18 and 70 years of age, diurnally active
3. A history of asthma diagnosed by physician at least 3 months prior to Visit 1 at GINA treatment steps 3 or 4. The diagnosis of asthma must have been made before the age of 40.
4. Pre-bronchodilator FEV1 between 60% predicted and 90% predicted at Visit 1.
5. Increase in FEV1 greater or equal to 12% and 200 ml 15 minutes after 400mcg salbutamol (albuterol) at Visit 1.
6. Patient must have been taking inhaled corticosteroids (ICS) for at least 12 weeks prior to screening, and must have been receiving at a stable dose for at least 6 weeks prior to screening either: - a medium to high dose ICS or - a low to high dose ICS in combination with Long acting beta agonist (LABA).
7. All patients must be symptomatic.

Exclusion criteria:

1. Patients with a significant disease other than asthma; a significant disease is defined as a disease which, in the opinion of the investigator, may (i) put the patient at risk because of participation in the study, (ii) influence the results of the study, or (iii) cause concern regarding the patient's ability to participate in the study
2. Patients who have been hospitalised for an asthma exacerbation within 3 months or had an admission to an intensive care unit for asthma within 3 years of Visit 1
3. Patients will be excluded when they have: - an aspartate aminotransferase (AST) >80 IU/L, alanine aminotransferase (ALT) >80 IU/L, bilirubin >1.5 X upper limit of normal (ULN) or creatinine >1.5 X ULN - clinically relevant abnormal baseline haematology, blood chemistry, or urinalysis
4. Patients with any of the following conditions: - a diagnosis of thyrotoxicosis

   * a diagnosis of paroxysmal tachycardia (>100 beats per minute)
   * a marked baseline prolongation of QT/QTc interval at Visit 1 (e.g., repeated demonstration of a QTc interval >450 ms) as recommended by ICH E14
   * a history of additional risk factors for Torsade de Pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome) as recommended by ICH E14.
5. Patients with any of the following conditions: - a history of myocardial infarction within 1 year of screening visit (Visit 1)

   * a diagnosis of clinically relevant cardiac arrhythmia
   * a history of cor pulmonale
   * known active tuberculosis
   * a malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years (patients with treated basal cell carcinoma are allowed)
   * a history of life-threatening pulmonary obstruction
   * a history of chronic obstructive pulmonary disease
   * history of cystic fibrosis
   * clinically evident bronchiectasis
   * a history of significant alcohol or drug abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2010-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (27):
- Austria (4):
  - 1222.27.43002 Boehringer Ingelheim Investigational Site, Linz
  - 1222.27.43004 Boehringer Ingelheim Investigational Site, Schlüsslberg
  - 1222.27.43001 Boehringer Ingelheim Investigational Site, Thalheim bei Wels
  - 1222.27.43003 Boehringer Ingelheim Investigational Site, Vienna
- Germany (9):
  - 1222.27.49003 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.27.49004 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.27.49009 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.27.49011 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1222.27.49008 Boehringer Ingelheim Investigational Site, Hanover
  - 1222.27.49002 Boehringer Ingelheim Investigational Site, Lübeck
  - 1222.27.49007 Boehringer Ingelheim Investigational Site, Rüdersdorf
  - 1222.27.49006 Boehringer Ingelheim Investigational Site, Wiesbaden
  - 1222.27.49010 Boehringer Ingelheim Investigational Site, Wiesloch
- Poland (4):
  - 1222.27.48001 Boehringer Ingelheim Investigational Site, Lodz
  - 1222.27.48002 Boehringer Ingelheim Investigational Site, Lodz
  - 1222.27.48003 Boehringer Ingelheim Investigational Site, Poznan
  - 1222.27.48004 Boehringer Ingelheim Investigational Site, Proszowice
- Romania (2):
  - 1222.27.40002 Boehringer Ingelheim Investigational Site, Bucharest
  - 1222.27.40003 Boehringer Ingelheim Investigational Site, Bucharest
- Slovakia (4):
  - 1222.27.42101 Boehringer Ingelheim Investigational Site, Bardejov
  - 1222.27.42103 Boehringer Ingelheim Investigational Site, Lučenec
  - 1222.27.42104 Boehringer Ingelheim Investigational Site, Martin
  - 1222.27.42102 Boehringer Ingelheim Investigational Site, Spišská Nová Ves
- Slovenia (4):
  - 1222.27.38601 Boehringer Ingelheim Investigational Site, Golnik
  - 1222.27.38605 Boehringer Ingelheim Investigational Site, Kamnik
  - 1222.27.38604 Boehringer Ingelheim Investigational Site, Topolšica
  - 1222.27.38603 Boehringer Ingelheim Investigational Site, Zgornje Hoče

REFERENCES:
- [Derived] O'Byrne PM, D'Urzo T, Beck E, Flezar M, Gahlemann M, Hart L, Blahova Z, Toorawa R, Beeh KM. Dose-finding evaluation of once-daily treatment with olodaterol, a novel long-acting beta2-agonist, in patients with asthma: results of a parallel-group study and a crossover study. Respir Res. 2015 Aug 18;16(1):97. doi: 10.1186/s12931-015-0249-8. PMID 26283085

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Total: This was a randomised, double-blind, double dummy, placebo- and active-controlled, 6 treatment, 4 period incomplete crossover trial. 198 patients were assigned randomly to one of 30 treatment sequences, each sequence comprising 4 out of the 6 treatments listed: one of four doses (20 microgram (mcg), 10 mcg, 5 mcg or 2 mcg) of Olodaterol (Olo) once daily (qd) delivered via the Respimat inhaler or Foradil (Form) 12 mcg twice daily (bid) delivered via the Aerolizer inhaler or equivalent placebo. The duration of each treatment period was 4 weeks with no washout periods between treatments.
Period: Overall Study
Arm/Group | Study Total
Started | 198 (Entered and treated)
Received Placebo | 125
Received Olo 2 mcg qd | 121
Received Olo 5 mcg qd | 130
Received Olo 10 mcg qd | 127
Received Olo 20 mcg qd | 124
Received Form 12 mcg Bid | 125
Completed | 182
Not Completed | 16
Not completed — Adverse Event | 8
Not completed — Protocol Violation | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | Study Total
Number analyzed (Participants) | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112
  Male | 86

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-24 Hours (AUC 0-24h) Response at the End of Each Treatment Period
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values at the randomisation visit. Means are adjusted for treatment, period, patient and study baseline. FEV1 AUC 0-24h was calculated from 0-24 hours post-dose using the trapezoidal rule, divided by the observation time (24h) to report in litres.
Time Frame: 1 hour (h) prior and 10 minutes (min) prior to first dose (baseline) and -1 h, -10 mins, 30 min, 60 min, 2 h, 3 h, 4 h, 11 h 50 min, 12 h 30 min, 13 h, 14 h, 15 h, 16 h, 18 h, 20 h, 22 h, 23 h, and 23 h 50 min related to evening dose after 4 weeks
Population: Full analysis set (FAS). FAS is defined as all patients in the treated set for whom the baseline (pre-dose) value is available, and who have a value for the primary endpoint for at least one crossover period.
Measure: Mean (Standard Error); unit: Liter
Groups:
- Placebo: Equivalent Placebo (morning and evening) delivered by the matching Inhaler (Respimat or Aerolizer).
- Olo 2 mcg qd: Olodaterol 2 mcg qd (evening, equivalent placebo morning) delivered by the Respimat Inhaler.
- Olo 5 mcg qd: Olodaterol 5 mcg qd (evening, equivalent placebo morning) delivered by the Respimat Inhaler.
- Olo 10 mcg qd: Olodaterol 10 mcg qd (evening, equivalent placebo morning) delivered by the Respimat Inhaler.
- Olo 20 mcg qd: Olodaterol 20 mcg qd (evening, equivalent placebo morning) delivered by the Respimat Inhaler.
- Form 12 mcg Bid: Foradil 12 mcg bid (morning and evening) delivered by the Aerolizer Inhaler.
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 121 | 119 | 122
Liter | -0.004 (0.025) | 0.135 (0.025) | 0.178 (0.025) | 0.201 (0.025) | 0.225 (0.025) | 0.164 (0.025)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted using a mixed model with treatment, period and study baseline value as fixed effects; and patients as random effect; Mean Difference (Final Values) = 0.140, 95% CI [0.097 to 0.182], Standard Error of Mean 0.022 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.182, 95% CI [0.140 to 0.224], Standard Error of Mean 0.021 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.205, 95% CI [0.163 to 0.248], Standard Error of Mean 0.022 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.229, 95% CI [0.186 to 0.272], Standard Error of Mean 0.022 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.169, 95% CI [0.126 to 0.211], Standard Error of Mean 0.022 — Form 12 mcg bid minus Placebo

2. Secondary Outcome: FEV1 Area Under Curve 0-12 h (AUC 0-12h) Response at the End of Each Treatment Period
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values at the randomisation visit. Means are adjusted for treatment, period, patient and study baseline. FEV1 AUC 0-12h was calculated from 0-12 hours post-dose using the trapezoidal rule, divided by the observation time (12h) to report in litres.
Time Frame: 1 hour (h) prior and 10 minutes (min) prior to first dose (baseline) and -1 h, -10 mins, 30 min, 60 min, 2 h, 3 h, 4 h, 11 h 50 min related to evening dose after 4 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 121 | 119 | 122
Liter | -0.039 (0.026) | 0.124 (0.026) | 0.173 (0.026) | 0.194 (0.026) | 0.211 (0.026) | 0.145 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.163, 95% CI [0.116 to 0.211], Standard Error of Mean 0.024 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.212, 95% CI [0.166 to 0.259], Standard Error of Mean 0.024 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.233, 95% CI [0.186 to 0.280], Standard Error of Mean 0.024 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.250, 95% CI [0.203 to 0.298], Standard Error of Mean 0.024 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.184, 95% CI [0.137 to 0.231], Standard Error of Mean 0.024 — Form 12 mcg bid minus Placebo

3. Secondary Outcome: FEV1 Area Under Curve 12-24 h (AUC 12-24h) Response at the End of Each Treatment Period
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values at the randomisation visit. Means are adjusted for treatment, period, patient and study baseline. FEV1 AUC 12-24h was calculated from 12-24 hours post-dose using the trapezoidal rule, divided by the observation time (12h) to report in litres.
Time Frame: 1 hour (h) prior and 10 minutes (min) prior to first dose (baseline) and 11 h 50 min, 12 h 30 min, 13 h, 14 h, 15 h, 16 h, 18 h, 20 h, 22 h, 23 h, and 23 h 50 min related to evening dose after 4 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 121 | 119 | 122
Liter | 0.031 (0.026) | 0.147 (0.026) | 0.183 (0.025) | 0.208 (0.026) | 0.238 (0.026) | 0.183 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.115, 95% CI [0.073 to 0.158], Standard Error of Mean 0.022 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.151, 95% CI [0.110 to 0.193], Standard Error of Mean 0.021 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.177, 95% CI [0.135 to 0.219], Standard Error of Mean 0.022 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.207, 95% CI [0.164 to 0.250], Standard Error of Mean 0.022 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.152, 95% CI [0.110 to 0.194], Standard Error of Mean 0.022 — Form 12 mcg bid minus Placebo

4. Secondary Outcome: Peak FEV1 Within 24 Hours Post-dose Response
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values at the randomisation visit. Peak FEV1 within 24 hours post dose measured following the evening trial drug inhalation at the end of each 4 week period of randomised treatment. Means are adjusted for treatment, period, patient and study baseline.
Time Frame: 1 hour (h) prior and 10 minutes (min) prior to first dose (baseline) and 30 min, 60 min, 2 h, 3 h, 4 h, 11 h 50 min, 12 h 30 min, 13 h, 14 h, 15 h, 16 h, 18 h, 20 h, 22 h, 23 h, and 23 h 50 min related to evening dose after 4 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 121 | 119 | 122
Liter | 0.224 (0.026) | 0.326 (0.027) | 0.359 (0.026) | 0.385 (0.027) | 0.404 (0.027) | 0.390 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.102, 95% CI [0.056 to 0.148], Standard Error of Mean 0.023 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.135, 95% CI [0.090 to 0.180], Standard Error of Mean 0.023 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.161, 95% CI [0.116 to 0.207], Standard Error of Mean 0.023 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.180, 95% CI [0.134 to 0.226], Standard Error of Mean 0.023 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.166, 95% CI [0.120 to 0.211], Standard Error of Mean 0.023 — Form 12 mcg bid minus Placebo

5. Secondary Outcome: Trough FEV1 Response
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values at the randomisation visit. Trough values were defined as the mean of 2 FEV1 values performed at the planned timepoints 23h and 23h 50min related to evening trial-drug inhalation at the end of each 4 week period of randomised treatment. Means are adjusted for treatment, period, patient and study baseline.
Time Frame: 1 hour (h) prior and 10 minutes (min) prior to first dose (baseline) and 23 h, and 23 h 50 min related to evening dose after 4 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 121 | 119 | 122
Liter | 0.013 (0.026) | 0.116 (0.026) | 0.146 (0.026) | 0.182 (0.026) | 0.211 (0.026) | 0.115 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.103, 95% CI [0.058 to 0.148], Standard Error of Mean 0.023 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.133, 95% CI [0.088 to 0.177], Standard Error of Mean 0.023 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.169, 95% CI [0.124 to 0.214], Standard Error of Mean 0.023 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.199, 95% CI [0.153 to 0.244], Standard Error of Mean 0.023 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.103, 95% CI [0.058 to 0.147], Standard Error of Mean 0.023 — Form 12 mcg bid minus Placebo

6. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-12 Hours (AUC 0-12h) Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values at the randomisation visit. Means are adjusted for treatment, period, patient and study baseline. FVC AUC 0-12h was calculated using the trapezoidal rule, divided by the observation time to report in litres.
Time Frame: 1 hour (h) prior and 10 minutes (min) prior to first dose (baseline) and -1 h, -10 mins, 30 min, 60 min, 2 h , 3 h, 4 h, 11 h 50 min related to evening dose after 4 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 121 | 119 | 122
Liter | -0.047 (0.029) | 0.056 (0.029) | 0.109 (0.029) | 0.094 (0.029) | 0.122 (0.029) | 0.055 (0.029)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.103, 95% CI [0.052 to 0.154], Standard Error of Mean 0.026 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.156, 95% CI [0.106 to 0.207], Standard Error of Mean 0.026 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.141, 95% CI [0.091 to 0.192], Standard Error of Mean 0.026 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.169, 95% CI [0.118 to 0.221], Standard Error of Mean 0.026 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.102, 95% CI [0.051 to 0.153], Standard Error of Mean 0.026 — Form 12 mcg bid minus Placebo

7. Secondary Outcome: FVC Area Under Curve 12-24 Hours (AUC 12-24h) Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values at the randomisation visit. Means are adjusted for treatment, period, patient and study baseline. FVC AUC 12-24h was calculated using the trapezoidal rule, divided by the observation time to report in litres.
Time Frame: as for outcome 3
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 121 | 119 | 122
Liter | -0.005 (0.029) | 0.055 (0.029) | 0.109 (0.028) | 0.110 (0.029) | 0.139 (0.029) | 0.085 (0.029)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0107, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.061, 95% CI [0.014 to 0.107], Standard Error of Mean 0.024 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.115, 95% CI [0.069 to 0.160], Standard Error of Mean 0.023 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.115, 95% CI [0.069 to 0.161], Standard Error of Mean 0.024 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.144, 95% CI [0.098 to 0.191], Standard Error of Mean 0.024 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.091, 95% CI [0.044 to 0.137], Standard Error of Mean 0.024 — Form 12 mcg bid minus Placebo

8. Secondary Outcome: FVC Area Under Curve 0-24 Hours (AUC 0-24h) Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values at the randomisation visit. Means are adjusted for treatment, period, patient and study baseline. FVC AUC 0-24h was calculated using the trapezoidal rule, divided by the observation time to report in litres.
Time Frame: 1 hour (h) prior and 10 minutes (min) prior to first dose (baseline) and -1 h, -10 min, 30 min, 60 min, 2 h, 3 h, 4 h, 11 h 50 min, 12 h 30 min, 13 h, 14 h, 15 h, 16 h, 18 h, 20 h, 22 h, 23 h, and 23 h 50 min related to evening dose after 4 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 121 | 119 | 122
Liter | -0.026 (0.028) | 0.056 (0.028) | 0.109 (0.028) | 0.102 (0.028) | 0.131 (0.028) | 0.070 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.082, 95% CI [0.036 to 0.128], Standard Error of Mean 0.023 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.136, 95% CI [0.090 to 0.181], Standard Error of Mean 0.023 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.128, 95% CI [0.083 to 0.174], Standard Error of Mean 0.023 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.157, 95% CI [0.111 to 0.203], Standard Error of Mean 0.023 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.097, 95% CI [0.051 to 0.143], Standard Error of Mean 0.023 — Form 12 mcg bid minus Placebo

9. Secondary Outcome: Peak FVC Within 24 Hours Post-dose Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values at the randomisation visit. Peak FVC within 24 hours post dose measured following the trial drug inhalation at the end of each 4 week period of randomised treatment. Means are adjusted for treatment, period, patient and study baseline.
Time Frame: as for outcome 4
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 121 | 119 | 122
Liter | 0.253 (0.031) | 0.300 (0.031) | 0.356 (0.031) | 0.342 (0.031) | 0.380 (0.031) | 0.326 (0.031)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0952, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.048, 95% CI [-0.008 to 0.103], Standard Error of Mean 0.028 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.103, 95% CI [0.048 to 0.158], Standard Error of Mean 0.028 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0016, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.089, 95% CI [0.034 to 0.145], Standard Error of Mean 0.028 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.127, 95% CI [0.071 to 0.183], Standard Error of Mean 0.028 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p = 0.0096, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.073, 95% CI [0.018 to 0.129], Standard Error of Mean 0.028 — Form 12 mcg bid minus Placebo

10. Secondary Outcome: Trough FVC Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values at the randomisation visit. Trough values were defined as the mean of 2 FEV1 values performed at the planned timepoints 23h and 23h 50min related to evening trial-drug inhalation at the end of each 4 week period of randomised treatment. Means are adjusted for treatment, period, patient and study baseline.
Time Frame: as for outcome 5
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 121 | 119 | 122
Liter | -0.022 (0.029) | 0.015 (0.029) | 0.069 (0.029) | 0.088 (0.029) | 0.107 (0.029) | 0.029 (0.029)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.1470, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.037, 95% CI [-0.013 to 0.088], Standard Error of Mean 0.026 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.091, 95% CI [0.042 to 0.141], Standard Error of Mean 0.025 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.110, 95% CI [0.060 to 0.160], Standard Error of Mean 0.025 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.129, 95% CI [0.078 to 0.179], Standard Error of Mean 0.026 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p = 0.0448, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.051, 95% CI [0.001 to 0.101], Standard Error of Mean 0.025 — Form 12 mcg bid minus Placebo

11. Secondary Outcome: Peak Expiratory Flow (PEF) Area Under Curve 0-12 Hours (AUC 0-12h) Response
Description: Response was defined as change from baseline. Study baseline PEF was defined as the mean of the available pre-dose PEF values at the randomisation visit. Means are adjusted for treatment, period, patient and study baseline. PEF AUC 0-12h was calculated using the trapezoidal rule, divided by the observation time to report in litres/seconds.
Time Frame: as for outcome 2
Population: FAS
Measure: Mean (Standard Error); unit: Liter/sec
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 121 | 119 | 122
Liter/sec | -0.117 (0.076) | 0.291 (0.077) | 0.449 (0.076) | 0.495 (0.077) | 0.553 (0.077) | 0.471 (0.076)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.408, 95% CI [0.277 to 0.539], Standard Error of Mean 0.067 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.566, 95% CI [0.438 to 0.695], Standard Error of Mean 0.066 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.612, 95% CI [0.482 to 0.743], Standard Error of Mean 0.066 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.670, 95% CI [0.539 to 0.801], Standard Error of Mean 0.067 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.588, 95% CI [0.457 to 0.718], Standard Error of Mean 0.066 — Form 12 mcg bid minus Placebo

12. Secondary Outcome: PEF Area Under Curve 12-24 Hours (AUC 12-24h) Response
Description: Response was defined as change from baseline. Study baseline PEF was defined as the mean of the available pre-dose PEF values at the randomisation visit. Means are adjusted for treatment, period, patient and study baseline. PEF AUC 12-24h was calculated using the trapezoidal rule, divided by the observation time to report in litres/seconds.
Time Frame: as for outcome 3
Population: FAS
Measure: Mean (Standard Error); unit: Liter/sec
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 121 | 119 | 122
Liter/sec | 0.043 (0.075) | 0.380 (0.075) | 0.528 (0.075) | 0.575 (0.075) | 0.692 (0.075) | 0.594 (0.075)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.337, 95% CI [0.213 to 0.461], Standard Error of Mean 0.063 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.485, 95% CI [0.363 to 0.606], Standard Error of Mean 0.062 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.531, 95% CI [0.408 to 0.655], Standard Error of Mean 0.063 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.648, 95% CI [0.524 to 0.772], Standard Error of Mean 0.063 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.551, 95% CI [0.428 to 0.674], Standard Error of Mean 0.063 — Form 12 mcg bid minus Placebo

13. Secondary Outcome: Peak Expiratory Flow (PEF) Area Under Curve 0-24 Hours (AUC 0-24h) Response
Description: Response was defined as change from baseline. Study baseline PEF was defined as the mean of the available pre-dose PEF values at the randomisation visit. Means are adjusted for treatment, period, patient and study baseline. PEF AUC 0-24h was calculated using the trapezoidal rule, divided by the observation time to report in litres/seconds.
Time Frame: 1 hour (h) prior and 10 minutes (min) prior to first dose (baseline) and -1h, -10 mins, 30 min, 60 min, 2 h, 3 h, 4 h, 11 h 50 min, 12 h 30 min, 13 h, 14 h, 15 h, 16 h, 18 h, 20 h, 22 h, 23 h, and 23 h 50 min related to evening dose after 4 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter/sec
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 121 | 119 | 122
Liter/sec | -0.038 (0.074) | 0.336 (0.074) | 0.489 (0.074) | 0.534 (0.074) | 0.623 (0.074) | 0.532 (0.074)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.373, 95% CI [0.253 to 0.493], Standard Error of Mean 0.061 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.527, 95% CI [0.409 to 0.645], Standard Error of Mean 0.060 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.572, 95% CI [0.453 to 0.692], Standard Error of Mean 0.061 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.660, 95% CI [0.540 to 0.781], Standard Error of Mean 0.061 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.570, 95% CI [0.451 to 0.689], Standard Error of Mean 0.061 — Form 12 mcg bid minus Placebo

14. Secondary Outcome: Peak PEF Within 24 Hours Post-dose Response
Description: Response was defined as change from baseline. Study baseline PEF was defined as the mean of the available pre-dose PEF values at the randomisation visit. Peak PEF within 24 hours post-dose measured following the evening trial drug inhalation at the end of each 4 week period of randomised treatment. Means are adjusted for treatment, period, patient and study baseline.
Time Frame: as for outcome 4
Population: FAS
Measure: Mean (Standard Error); unit: Liter/sec
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 121 | 119 | 122
Liter/sec | 0.664 (0.079) | 0.966 (0.079) | 1.093 (0.078) | 1.130 (0.079) | 1.198 (0.079) | 1.168 (0.079)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.302, 95% CI [0.168 to 0.436], Standard Error of Mean 0.068 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.429, 95% CI [0.297 to 0.561], Standard Error of Mean 0.067 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.466, 95% CI [0.333 to 0.599], Standard Error of Mean 0.068 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.534, 95% CI [0.400 to 0.669], Standard Error of Mean 0.068 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.504, 95% CI [0.371 to 0.637], Standard Error of Mean 0.068 — Form 12 mcg bid minus Placebo

15. Secondary Outcome: Trough PEF Response
Description: Response was defined as change from baseline. Study baseline PEF was defined as the mean of the available pre-dose PEF values at the randomisation visit. Trough values were defined as the mean of 2 FEV1 values performed at the planned timepoints 23h and 23h 50min related to evening trial-drug inhalation at the end of each 4 week period of randomised treatment. Means are adjusted for treatment, period, patient and study baseline.
Time Frame: as for outcome 5
Population: FAS
Measure: Mean (Standard Error); unit: Liter/sec
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 121 | 119 | 122
Liter/sec | 0.031 (0.078) | 0.295 (0.078) | 0.499 (0.077) | 0.515 (0.078) | 0.655 (0.078) | 0.478 (0.078)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.264, 95% CI [0.127 to 0.401], Standard Error of Mean 0.070 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.468, 95% CI [0.333 to 0.602], Standard Error of Mean 0.069 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.484, 95% CI [0.348 to 0.620], Standard Error of Mean 0.069 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.624, 95% CI [0.487 to 0.761], Standard Error of Mean 0.070 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.447, 95% CI [0.311 to 0.583], Standard Error of Mean 0.069 — Form 12 mcg bid minus Placebo

16. Secondary Outcome: Mean Pre-dose Morning PEF (PEF a.m.)
Description: PEF a.m. was measured by patients at home using the AM2+ device (overall means obtained during each period of randomised treatment excluding the data of the first 2 weeks will be compared). Means are adjusted for treatment, period, patient and study baseline.
Time Frame: 2-4 weeks
Population: FAS including all patients who contributed data for this endpoint.
Measure: Mean (Standard Error); unit: Liter/min
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 123 | 120 | 123
Liter/min | 361.89 (4.548) | 383.90 (4.567) | 390.91 (4.519) | 389.78 (4.539) | 394.82 (4.560) | 385.42 (4.539)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 22.012, 95% CI [14.802 to 29.223], Standard Error of Mean 3.671 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 29.022, 95% CI [21.931 to 36.114], Standard Error of Mean 3.610 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 27.887, 95% CI [20.755 to 35.019], Standard Error of Mean 3.631 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 32.935, 95% CI [25.730 to 40.139], Standard Error of Mean 3.668 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 23.528, 95% CI [16.371 to 30.686], Standard Error of Mean 3.644 — Form 12 mcg bid minus Placebo

17. Secondary Outcome: Mean Pre-dose Evening PEF (PEF p.m.)
Description: PEF p.m. was measured by patients at home using the AM2+ device (overall means obtained during each period of randomised treatment excluding the data of the first 2 weeks will be compared). Means are adjusted for treatment, period, patient and study baseline.
Time Frame: 2-4 weeks
Population: FAS including all patients who contributed data for this endpoint.
Measure: Mean (Standard Error); unit: Liter/min
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 123 | 120 | 123
Liter/min | 379.44 (4.398) | 394.36 (4.418) | 404.28 (4.368) | 403.06 (4.389) | 407.89 (4.410) | 399.88 (4.389)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 14.920, 95% CI [7.770 to 22.071], Standard Error of Mean 3.640 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 24.834, 95% CI [17.801 to 31.866], Standard Error of Mean 3.580 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 23.613, 95% CI [16.539 to 30.686], Standard Error of Mean 3.601 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 28.449, 95% CI [21.305 to 35.594], Standard Error of Mean 3.637 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 20.439, 95% CI [13.341 to 27.538], Standard Error of Mean 3.614 — Form 12 mcg bid minus Placebo

18. Secondary Outcome: PEF Daily Variability
Description: PEF daily variability was assessed by patients at home using the AM2+ device (overall means obtained during each period of randomised treatment excluding the data of the first 2 weeks will be compared). PEF daily variability is the absolute difference between the morning and the evening PEF value divided by the mean of these two values, expressed as a percent. Means are adjusted for treatment, period, patient and study baseline.
Time Frame: 2-4 weeks
Population: FAS including all patients who contributed data for this endpoint.
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 122 | 120 | 123
Percentage | 11.688 (0.480) | 9.694 (0.484) | 9.593 (0.475) | 9.851 (0.480) | 9.899 (0.483) | 10.417 (0.479)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.994, 95% CI [-2.989 to -0.999], Standard Error of Mean 0.507 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.095, 95% CI [-3.073 to -1.116], Standard Error of Mean 0.498 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.836, 95% CI [-2.824 to -0.849], Standard Error of Mean 0.503 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.789, 95% CI [-2.783 to -0.795], Standard Error of Mean 0.506 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p = 0.0118, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.270, 95% CI [-2.258 to -0.283], Standard Error of Mean 0.503 — Form 12 mcg bid minus Placebo

19. Secondary Outcome: Mean Pre-dose Morning FEV1 (FEV1 a.m.)
Description: FEV1 a.m. was measured by patients at home using the AM2+ device (overall means obtained during each period of randomised treatment excluding the data of the first 2 weeks will be compared). Means are adjusted for treatment, period, patient and study baseline.
Time Frame: 2-4 weeks
Population: FAS including all patients who contributed data for this endpoint.
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 123 | 120 | 123
L | 2.309 (0.028) | 2.402 (0.028) | 2.438 (0.028) | 2.445 (0.028) | 2.479 (0.028) | 2.403 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.093, 95% CI [0.045 to 0.141], Standard Error of Mean 0.025 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.128, 95% CI [0.081 to 0.176], Standard Error of Mean 0.024 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.135, 95% CI [0.087 to 0.183], Standard Error of Mean 0.024 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.169, 95% CI [0.121 to 0.217], Standard Error of Mean 0.025 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.093, 95% CI [0.045 to 0.141], Standard Error of Mean 0.024 — Form 12 mcg bid minus Placebo

20. Secondary Outcome: Mean Pre-dose Evening FEV1 (FEV1 p.m.)
Description: FEV1 p.m. was measured by patients at home using the AM2+ device (overall means obtained during each period of randomised treatment excluding the data of the first 2 weeks will be compared). Means are adjusted for treatment, period, patient and study baseline.
Time Frame: 2-4 weeks
Population: FAS including all patients who contributed data for this endpoint.
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 123 | 120 | 123
L | 2.378 (0.027) | 2.428 (0.027) | 2.460 (0.027) | 2.467 (0.027) | 2.495 (0.027) | 2.457 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0362, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.050, 95% CI [0.003 to 0.097], Standard Error of Mean 0.024 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.081, 95% CI [0.035 to 0.127], Standard Error of Mean 0.023 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.088, 95% CI [0.042 to 0.135], Standard Error of Mean 0.024 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.117, 95% CI [0.070 to 0.164], Standard Error of Mean 0.024 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p = 0.0010, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.079, 95% CI [0.032 to 0.125], Standard Error of Mean 0.024 — Form 12 mcg bid minus Placebo

21. Secondary Outcome: Mean Number of Puffs of Rescue Medication During the Whole Day
Description: Mean of daily use of salbutamol (albuterol) rescue medication as needed during the entire study period. Assessed by patients at home using the AM2+ device (overall means obtained during each period of randomised treatment excluding the data of the first 2 weeks will be compared). Means are adjusted for treatment, period, patient and study baseline.
Time Frame: 2-4 weeks
Population: FAS including all patients who contributed data for this endpoint.
Measure: Mean (Standard Error); unit: Number of Puffs
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 123 | 120 | 123
Number of Puffs | 1.749 (0.130) | 1.222 (0.130) | 1.317 (0.128) | 1.271 (0.129) | 1.092 (0.130) | 1.300 (0.129)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.526, 95% CI [-0.770 to -0.282], Standard Error of Mean 0.124 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.432, 95% CI [-0.671 to -0.192], Standard Error of Mean 0.122 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.478, 95% CI [-0.720 to -0.237], Standard Error of Mean 0.123 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.657, 95% CI [-0.901 to -0.413], Standard Error of Mean 0.124 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.449, 95% CI [-0.691 to -0.207], Standard Error of Mean 0.123 — Form 12 mcg bid minus Placebo

22. Secondary Outcome: Percentage of Asthma Symptom Free Days
Description: Percentage of asthma-symptom free days after the first 2 weeks of each treatment period was calculated as the number of symptom-free days divided by the number of days on treatment multiplied by 100. A symptom-free day was defined as a day in which no asthma symptoms were recorded, no rescue medication was recorded, activities during the day were not at all limited due to asthma, no shortness of breath during the day was recorded, no wheezing or coughing during the day and no night-time awakenings due to asthma were recorded. Assessed by patients at home using the AM2+ device.
Time Frame: 2-4 weeks
Population: FAS including all patients who contributed data for this endpoint.
Measure: Mean (Standard Error); unit: Percentage of asthma symptom free days
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 123 | 119 | 126 | 123 | 120 | 123
Percentage of asthma symptom free days | 18.502 (2.494) | 26.430 (2.973) | 22.348 (2.835) | 23.624 (2.951) | 21.326 (2.803) | 23.664 (2.797)

23. Secondary Outcome: Number of Patients Categorized by Highest Number of Night Time Awakenings (Overall)
Description: Assessed by patients at home using the AM2+ device after the first 2 weeks of each period of randomised treatment.
Time Frame: 2-4 weeks
Population: FAS including all patients who contributed data for this endpoint.
Measure: Number; unit: Number of patients
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 123 | 120 | 123
Number of patients
  Did not wake up | 55 | 60 | 58 | 56 | 63 | 59
  Woke up once | 37 | 36 | 34 | 34 | 34 | 29
  Woke up 2-5 times | 26 | 17 | 30 | 30 | 20 | 33
  Woke up > 5 times | 3 | 5 | 2 | 1 | 2 | 2
  Was awake all night | 1 | 1 | 2 | 2 | 1 | 0

24. Secondary Outcome: Number of Patients Categorized by Worst Asthma Daytime Symptoms (Overall)
Description: Assessed by patients at home using the AM2+ device after the first 2 weeks of each period of randomised treatment.
Time Frame: 2-4 weeks
Population: FAS including all patients who contributed data for this endpoint.
Measure: Number; unit: Number of patients
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 123 | 120 | 123
Number of patients
  No asthma symptoms | 20 | 26 | 29 | 23 | 21 | 24
  Mild asthma symptoms | 31 | 46 | 29 | 37 | 38 | 37
  Moderate asthma symptoms | 56 | 37 | 51 | 52 | 54 | 49
  Severe asthma symptoms | 15 | 10 | 12 | 10 | 6 | 12
  Very severe asthma symptoms | 0 | 0 | 5 | 1 | 1 | 1

25. Secondary Outcome: Number of Patients Categorized by Worst Asthma Nighttime Symptoms (Overall)
Description: Assessed by patients at home using the AM2+ device after the first 2 weeks of each period of randomised treatment.
Time Frame: 2-4 weeks
Population: FAS including all patients who contributed data for this endpoint.
Measure: Number; unit: Number of patients
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 126 | 123 | 120 | 123
Number of patients
  No asthma symptoms | 27 | 31 | 22 | 25 | 27 | 26
  Mild asthma symptoms | 32 | 47 | 48 | 40 | 45 | 39
  Moderate asthma symptoms | 49 | 29 | 45 | 46 | 43 | 46
  Severe asthma symptoms | 14 | 10 | 11 | 10 | 5 | 10
  Very severe asthma symptoms | 0 | 2 | 0 | 2 | 0 | 2

26. Secondary Outcome: Total Asthma Quality of Life Questionnaire (AQLQ(s)) Score
Description: Total score from the Standardised Asthma Quality of Life Questionnaire (AQLQ (s)) at the end of each 4 week treatment period. The AQLQ(s) contains 32 questions, each question has a 7 point scale from 1 (highest intensity) till 7 (no symptoms). Total score was defined as the sum of all items divided by the number of items.
Time Frame: 4 weeks
Population: FAS including all patients who contributed data for this endpoint.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 122 | 119 | 125 | 121 | 118 | 122
units on a scale | 5.174 (0.063) | 5.463 (0.064) | 5.383 (0.063) | 5.437 (0.063) | 5.491 (0.064) | 5.489 (0.063)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.289, 95% CI [0.178 to 0.400], Standard Error of Mean 0.057 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.209, 95% CI [0.099 to 0.318], Standard Error of Mean 0.056 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.262, 95% CI [0.151 to 0.374], Standard Error of Mean 0.057 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.317, 95% CI [0.205 to 0.429], Standard Error of Mean 0.057 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.315, 95% CI [0.203 to 0.426], Standard Error of Mean 0.057 — Form 12 mcg bid minus Placebo

27. Secondary Outcome: Total Asthma Control Questionnaire (ACQ) Score
Description: Control of asthma as assessed by the ACQ at the end of each 4-week treatment period.The ACQ contains 7 questions, each question has a 7 point scale from 0 (no symptoms) till 6 (highest intensity). Total score was defined as the sum of all items divided by the number of items.
Time Frame: 4 weeks
Population: FAS including all patients who contributed data for this endpoint.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 123 | 119 | 126 | 122 | 119 | 122
units on a scale | 1.882 (0.058) | 1.561 (0.058) | 1.589 (0.057) | 1.556 (0.058) | 1.488 (0.058) | 1.536 (0.058)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.321, 95% CI [-0.432 to -0.210], Standard Error of Mean 0.057 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.293, 95% CI [-0.403 to -0.184], Standard Error of Mean 0.056 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.326, 95% CI [-0.436 to -0.215], Standard Error of Mean 0.056 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.394, 95% CI [-0.505 to -0.282], Standard Error of Mean 0.057 — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.346, 95% CI [-0.457 to -0.235], Standard Error of Mean 0.056 — Form 12 mcg bid minus Placebo

28. Secondary Outcome: Potassium 1 Hour Pre-dose
Description: Effect on potassium evaluated 1 hour pre-dose. Analysis is based on the log of the potassium values. For the geometric means, the results were back-transformed to the original scale.
Time Frame: 4 weeks
Population: Treated set
Measure: Geometric Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 119 | 118 | 122 | 117 | 117 | 119
mmol/L | 4.067 [4.019 to 4.114] | 4.051 [4.004 to 4.099] | 4.051 [4.005 to 4.097] | 4.061 [4.014 to 4.109] | 4.057 [4.010 to 4.105] | 4.080 [4.032 to 4.128]
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.6187, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 0.996, 95% CI [0.981 to 1.011] — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.6022, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 0.996, 95% CI [0.981 to 1.011] — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.8641, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 0.999, 95% CI [0.984 to 1.014] — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.7664, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 0.998, 95% CI [0.983 to 1.013] — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p = 0.6757, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 1.003, 95% CI [0.988 to 1.018] — Form 12 mcg bid minus Placebo

29. Secondary Outcome: Potassium 1 Hour Post-dose
Description: Effect on potassium evaluated 1 hour post-dose. Analysis is based on the log of the potassium values. For the geometric means, the results were back-transformed to the original scale.
Time Frame: 4 weeks
Population: Treated set
Measure: Geometric Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 115 | 113 | 118 | 114 | 109 | 114
mmol/L | 4.097 [4.040 to 4.155] | 4.069 [4.012 to 4.126] | 4.013 [3.958 to 4.069] | 4.004 [3.948 to 4.060] | 4.015 [3.957 to 4.073] | 4.059 [4.003 to 4.117]
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.4423, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 0.993, 95% CI [0.975 to 1.011] — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0218, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 0.979, 95% CI [0.962 to 0.997] — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0109, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 0.977, 95% CI [0.960 to 0.995] — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0283, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 0.980, 95% CI [0.962 to 0.998] — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p = 0.3085, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 0.991, 95% CI [0.973 to 1.009] — Form 12 mcg bid minus Placebo

30. Secondary Outcome: Potassium 3 Hours Post-dose
Description: Effect on potassium evaluated 3 hours post-dose. Analysis is based on the log of the potassium values. For the geometric means, the results were back-transformed to the original scale.
Time Frame: 4 weeks
Population: Treated set
Measure: Geometric Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 113 | 110 | 119 | 114 | 105 | 114
mmol/L | 4.029 [3.980 to 4.079] | 4.026 [3.976 to 4.076] | 3.997 [3.950 to 4.045] | 3.979 [3.931 to 4.027] | 3.992 [3.942 to 4.043] | 4.007 [3.959 to 4.056]
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.9112, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 0.999, 95% CI [0.984 to 1.015] — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.2955, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 0.992, 95% CI [0.977 to 1.007] — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.1029, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 0.987, 95% CI [0.973 to 1.003] — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.2552, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 0.991, 95% CI [0.975 to 1.007] — Olo 20 mcg qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p = 0.4803, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 0.994, 95% CI [0.979 to 1.010] — Form 12 mcg bid minus Placebo

31. Secondary Outcome: Clinical Relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis and ECG
Description: Clinical relevant abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis and ECG. New abnormal findings or worsening of baseline conditions were reported as Adverse Events.
Time Frame: 4 weeks
Population: Treated Set
Measure: Number; unit: Participants
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 125 | 121 | 130 | 127 | 124 | 125
Participants
  Atrioventricular block first degree | 0 | 0 | 0 | 0 | 1 | 1
  Blood creatine phosphokinase MB increased | 0 | 0 | 0 | 1 | 0 | 0
  Blood creatine phosphokinase increased | 0 | 0 | 0 | 1 | 0 | 0
  Blood pressure increased | 0 | 1 | 0 | 0 | 0 | 0
  Hypothyroidism | 0 | 0 | 1 | 0 | 0 | 0
  Hypertension | 0 | 0 | 1 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- Olo 2 mcg: Olodaterol 2 mcg qd (evening, equivalent placebo morning) delivered by the Respimat Inhaler.
- Olo 5 mcg: Olodaterol 5 mcg qd (evening, equivalent placebo morning) delivered by the Respimat Inhaler.
- Olo 10 mcg: Olodaterol 10 mcg qd (evening, equivalent placebo morning) delivered by the Respimat Inhaler.
- Olo 20 mcg: Olodaterol 20 mcg qd (evening, equivalent placebo morning) delivered by the Respimat Inhaler.
- Form 12 mcg: Foradil 12 mcg bid (morning and evening) delivered by the Aerolizer Inhaler.
Arm/Group | Placebo | Olo 2 mcg | Olo 5 mcg | Olo 10 mcg | Olo 20 mcg | Form 12 mcg
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/121 | 0/130 | 1/127 | 0/124 | 0/125
Other Adverse Events (participants affected / at risk) | 0/125 | 0/121 | 0/130 | 0/127 | 0/124 | 0/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=125) | Olo 2 mcg (N=121) | Olo 5 mcg (N=130) | Olo 10 mcg (N=127) | Olo 20 mcg (N=124) | Form 12 mcg (N=125)
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication